CLINICAL TRIAL: NCT04907006
Title: A Randomized, Open-label, Two-period, Double Crossover, Single Center Study to Evaluate the Effect of High-fat Diet on the Pharmacokinetics of SY-004 in Healthy Subjects
Brief Title: A Food-drug Interaction Study of SY-004 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SY004004
Record Dates: First submitted 2021-05-15; First posted 2021-05-28 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes
Keywords: Food drug interaction，Hypoglycemic drugs，SY-004
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-1 (Experimental): The subjects in both groups will be fasting overnight for at least 10 hours before administration. In Group-1 on D1, subjects will be orally administered with one SY-004 capsule(80mg ) on an empty stomach with 240ml warm water; In Group-2, subjects will have high-fat breakfast 30 minutes before administration ,then take one SY-004 capsule(80mg) orally with 240ml warm water.
  The subjects in both groups will be fasted within 4 hours after taking the medicine, and drinking water is forbidden within 1 hour before and after taking the medicine.
  After the cleaning period (D9-D16), the subjects will exchang the way of taking medicine and enter the second cycle of drug administration.
  Interventions: Drug: SY-004 capsule
- Group-2 (Experimental): The subjects in both groups will be fasting overnight for at least 10 hours before administration. In Group-1 on D1, subjects will be orally administered with one SY-004 capsule(80mg ) on an empty stomach with 240ml warm water; In Group-2, subjects will have high-fat breakfast 30 minutes before administration ,then take one SY-004 capsule(80mg) orally with 240ml warm water.
  The subjects in both groups will be fasted within 4 hours after taking the medicine, and drinking water is forbidden within 1 hour before and after taking the medicine.
  After the cleaning period (D9-D16), the subjects will exchang the way of taking medicine and enter the second cycle of drug administration.
  Interventions: Drug: SY-004 capsule

INTERVENTIONS:
Drug: SY-004 capsule — After fasting for 10 hours, subjects in group 1 took one SY-004 (80mg) orally on an empty stomach on the day of administration with 240ml warm water; Subjects in group 2 began to eat high-fat breakfast 30 minutes before administration , and took one SY-004 capsule（80mg） orally with 240ml warm water. The subjects in both groups were fasted within 4 hours after taking the medicine, and drinking water was forbidden within 1 hour before and after taking SY-004.

SUMMARY:
A randomized, open, two cycle, double crossover, single center study was conducted to evaluate the effect of high-fat diet on the pharmacokinetics of SY-004 in healthy subjects

DETAILED DESCRIPTION:
This study will evaluate the effect of high-fat diet on the pharmacokinetics of SY-004.

ELIGIBILITY:
Inclusion Criteria:

* The subjects can communicate well with the researchers, understand and comply with the requirements of this study, and sign the informed consent voluntarily.
* Age on the day of signing the informed consent: healthy subjects aged 18 or above, both male and female.
* At the time of screening, male weight ≥ 50.0 kg, female weight ≥ 45.0 kg, 19.0 kg / m2 ≤ BMI ≤ 26.0 kg / m2.
* Fasting blood glucose ≥ 3.9 mmol / L and < 6.1 mmol / L.
* From one month before the informed consent to three months after the last medication, the subjects and their partners had no plans to have a child, take effective contraceptive measures voluntarily, and donate sperm or eggs.

Exclusion Criteria:

* Within 3 months before screening, a clinical trial was completed or withdrawn, or a clinical trial was currently in progress, or other medical trials were conducted. The researchers judged that it was not suitable for the trial.
* In the past, there were serious systematic diseases or family history (including cardiovascular system, digestive system, urinary system, etc.), the researchers judged that the disease status could significantly change the absorption, distribution, metabolism and excretion of the drug used in the trial, or the risk of the subjects would be increased by taking the trial drug.
* Allergic constitution, or food allergy history, or known to be allergic to study drug / similar drug.
* Previous history of hypoglycemia.
* Previous patients with postural hypotension.
* The past five years have been positive for drug abuse, drug use history or urine drug screening results.
* Those who donate blood or lose more than 400ml of blood within 4 weeks before screening, or who have received blood or blood component infusion within 4 weeks before screening, or who plan to donate blood components within 3 months after the end of the study.
* Those who have history of syncope or blood sickness, who cannot tolerate venous puncture or have difficulty in blood collection.
* Severe infection, trauma or surgical operation within 4 weeks prior to screening, or those who are scheduled to perform surgery during the study (including, but not limited to, dental operations).
* Use any prescription, over-the-counter, herbal or health care product within 2 weeks prior to screening.
* Any drugs that inhibit or induce the metabolism of liver drugs were used within 30 days before screening.
* The average alcohol intake in the first three months of screening was more than 14 units per week (1 unit = 360ml beer, 45ml of alcohol content of 40% spirits or wine 150ml), or those who could not give up drinking alcohol during the test, or those who were positive for alcohol exhalation.
* Smoking was ≥ 5 cigarettes per day within 3 months before screening, or unwilling / unable to give up smoking during the trial.
* Special requirements for diet, and those who cannot comply with the unified diet arrangement.
* No guarantee of chocolate, any caffeine or food or drink (such as Firedragon fruit, grapefruit, grapefruit, orange juice, mango, etc.) 48 hours before and during the test.
* Pregnant or lactating women, or pregnant women with positive results.
* The results of screening were positive for HBsAg, HCV, TP and HIV.
* ALT > 1.5 times of normal value was found in screening（ × ULN), or glutamic transaminase (AST) >1.5 × ULN, or serum total bilirubin (TBIL) > 1.5 × ULN。
* The results of 12 lead ECG were: QT interval (qtcb) >450ms (male) or >470ms (female).
* The results of physical examination, vital signs, abdominal B-ultrasound (liver, gallbladder, pancreas, spleen and kidney), chest CT, ECG, laboratory examination items and related auxiliary examination results were judged by the researchers to be unsuitable for the participants.
* The researchers judged that the subjects with other factors were not suitable for participating in the test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
AUC0-t | 8 days
  Under fasting and high-fat diet, Area under the plasma concentration versus time curve (AUC) 0-t of SY-004 in human plasma.
AUC0-∞ | 8 days
  Under fasting and high-fat diet, Area under the plasma concentration versus time curve (AUC)0 - ∞ of SY-004 in human plasma.
Cmax | 8 days
  Under fasting and high-fat diet, Peak Plasma Concentration (Cmax) of SY-004 in human plasma.

SECONDARY OUTCOMES:
Tmax、t1/2z、CLz/F | 8 days
  Under fasting and high-fat diet, Peak time(Tmax) of SY-004 in human plasma.
t1/2z | 8 days
  Under fasting and high-fat diet, Half life (T1/2z) of SY-004 in human plasma.
CLz/F | 8 days
  Under fasting and high-fat diet, clearance (Cl) of SY-004 in human plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Haitang Xie, Dr, Principal Investigator — Wannan Medical College
Locations (1):
- XIE Haitang, Wuhu, Anhui, China